CLINICAL TRIAL: NCT03513003
Title: The Use of a Pacifier to Correct Malocclusions in Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZB-Pacifier
Record Dates: First submitted 2018-04-27; First posted 2018-05-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional pacifier (Experimental): Swap from the habitual pacifier to a functional pacifier
  Interventions: Device: Functional Pacifier
- Stop habit (Active Comparator): Stop the use of the habitual pacifier and or baby bottle
  Interventions: Behavioral: Stop habit

INTERVENTIONS:
Device: Functional Pacifier — Children swap from their habitual pacifier to the functional pacifier and stop baby bottle
  Arms: Functional pacifier
Behavioral: Stop habit — Children stop the use of their pacifier and/or baby bottle
  Arms: Stop habit

SUMMARY:
The aim of the study is to investigate the effect of a pacifier (102 Medical Pacifier, Curaprox, Switzerland) on malocclusions like posterior crossbite, anterior open bite, larger overjet and tongue dysfunction in young children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are sucking the pacifier and / or baby bottle for the last 6 months in use.
* Manifesting posterior crossbite in which minium 1 tooth and/or edge to edge in the region deciduous canines and/or deciduous molars, with or without forced bite.

AND / OR

- Manifesting anterior open bite in which the overbite has negative values or edge to edge (≤ 0), with or without tongue thrust.

Exclusion Criteria:

* Children who are thumb- or fingersucking (or sucking other objects)
* syndromic or cleft patients
* patients with history of cranio-facial trauma, history of temporomandibular joint infection or musculo-skeletal asymmetry (e.g. scoliosis, torticollis)
* patients with systematic diseases
* patients currently under or after orthodontic Treatment
* patients with ankylosed teeth (e.g. after dental trauma).

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Posterior cross bite | 1 year
  presence of posterior crossbite in which minium 1 tooth and/or edge to edge in the region deciduous canines and/or deciduous molars, with or without forced bite.
Anterior open bite | 1 year
  presence of anterior open bite in which the overbite has negative values or edge to edge (≤ 0), with or without tongue thrust.

SECONDARY OUTCOMES:
Facial movement | 1 year
  Lip contraction during swallowing of a sip of water
Lip competence | 1 year
  Contact between the upper and the lower lips at rest
Facial morphology | 1 year
  3D measurements of facial proportions

CONTACTS AND LOCATIONS:
Overall Officials: Carlalberta Verna, DDS, PhD, Study Chair — University Center for Dental Medicine, Basel, Switzerland
Locations (1):
- UZB, University Center for Dental Medicine, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimberg L, Bondemark L, Soderfeldt B, Lennartsson B. Prevalence of malocclusion traits and sucking habits among 3-year-old children. Swed Dent J. 2010;34(1):35-42. PMID 20496855
- [Background] Warren JJ, Slayton RL, Bishara SE, Levy SM, Yonezu T, Kanellis MJ. Effects of nonnutritive sucking habits on occlusal characteristics in the mixed dentition. Pediatr Dent. 2005 Nov-Dec;27(6):445-50. PMID 16532883
- [Background] Sousa RV, Pinto-Monteiro AK, Martins CC, Granville-Garcia AF, Paiva SM. Malocclusion and socioeconomic indicators in primary dentition. Braz Oral Res. 2014;28:54-60. doi: 10.1590/s1806-83242013005000032. PMID 25000602
- [Background] Filippi C, Filippi A, Verna C. [Orthodontic therapy in the early childhood using pacifier?]. Swiss Dent J. 2015;125(9):959-70. doi: 10.61872/sdj-2015-09-03. French, German. PMID 26399737
- [Background] Schmid KM, Kugler R, Nalabothu P, Bosch C, Verna C. The effect of pacifier sucking on orofacial structures: a systematic literature review. Prog Orthod. 2018 Mar 13;19(1):8. doi: 10.1186/s40510-018-0206-4. PMID 29532184